CLINICAL TRIAL: NCT07031011
Title: An Early Clinical Study to Investigate the Safety, Pharmacokinetics, and Efficacy of PD-1-M1-NK Cells (YC-T-001) in Patients With Advanced Gastric or Colorectal Cancer Failed or Intolerant to at Least Second-line Therapy
Brief Title: PD-1-M1-NK Cells in the Treatment of Advanced Gastric or Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: jiuwei cui (Other)
Responsible Party: Sponsor-Investigator, jiuwei cui, Chief Physician, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YC-T-001
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Advanced Gastric or Colorectal Cancer
Keywords: CAR-NK
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced gastric or colorectal cancer treated with PD-1-M1-CAR-NK Cells (YC-T-001) (Experimental): Subjects with advanced gastric cancer or colorectal cancer were treated with PD-1-M1-CAR-NK Cells (YC-T-001) in the form of intraperitoneal injection
  Interventions: Biological: PD-1-M1-NK Cells

INTERVENTIONS:
Biological: PD-1-M1-NK Cells — At dose escalation stage, four dose groups were initially determined: 5×106CAR NK cells/kg, 1×107CARNK cells/kg, 2×107CARNK cells/kg, and 5×107 CARNK cells/kg. Administration cycle: In Cycle 1 (C1), the drug was administered once on days 1, 4, 7, 10 and 13 respectively. A complete cycle was formed by five consecutive administrations. For subjects with stable, partial response or complete response in the tumor assessment at the first time in week 4, the treatment in Cycle 2 will continue subsequently. In Cycle 2, the drug was administered once every two weeks (Q2W: D14±7 days and D28±7 days).

SUMMARY:
This is an Early Clinical Study to Investigate the Safety, Pharmacokinetics, and Efficacy of PD-1-M1-NK Cells (YC-T-001) in Patients with Advanced Gastric or Colorectal Cancer Failed or Intolerant to at Least Second-line Therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited. Age should be between 18 and 75 years old (including the critical value), and one should be able to understand and voluntarily sign the informed consent form.
2. The ECOG performance status score is 0-1, and the expected survival period is no less than 3 months (judged by the researchers).
3. Advanced gastric cancer or colorectal cancer confirmed by histology, which has failed or been intolerant after at least two lines of standardized systematic treatment (including but not limited to targeted therapy, immunotherapy or chemotherapy), and has been confirmed as disease progression by imaging examination.
4. The subjects should be able to provide tumor tissue samples (archived tumor tissues within one year should be provided as much as possible) (at least 5-10 tumor tissue slices should be provided; if it is a surgical resection specimen, at least 10 slices should be provided). For patients in special circumstances who are unable to provide tissue samples or have less than 5 slices (or less than 10 surgical resection specimen slices), It is necessary to communicate with the partner to determine whether this selection criterion can be exempted. The tumor tissue samples were positive for PDL1+ by immunohistochemical detection.
5. There is at least one measurable lesion (in accordance with the RECIST 1.1 standard)
6. Unless otherwise specified, subjects should meet the following conditions before screening and pretreatment. If laboratory test abnormalities occur and do not meet the following standards, a re-examination within one week is allowed. If the standards are still not met, they will not be included:

   1. Blood routine test (no intensive blood transfusion (such as more than 2 blood transfations within 7 days), platelet transfusion, cell growth factor (except recombinant erythropoietin) and other supportive treatments within 7 days before the test) : Neutrophils (NE) ≥ 1.5×109/L, lymphocytes (LY) ≥ 0.4×109/L (except before pretreatment), platelets (PLT) ≥ 75×109/L, hemoglobin (Hb) ≥ 8.0 g/dL;
   2. Blood biochemistry: Endogenous creatinine clearance rate ≥ 50 mL/min (using the CockcrofT-GaulT formula), ALT ≤ 2.5×ULN, AST ≤ 2.5×ULN, total bilirubin ≤ 2×ULN; Serum lipase and amylase ≤ 1.5 ULN; Alkaline phosphatase ≤ 2.5 ULN; If bone or liver metastasis occurs, AST, ALT and alkaline phosphatase ≤ 5ULN;
   3. Prothrombin time (PT) ≤1.5×ULN; INR≤1.5×ULN; APTT≤1.5×ULN.
7. No active or uncontrolled central nervous system metastases (Patients with treated brain metastases who have stable symptoms and stable hormone doses for more than 4 weeks can be enrolled).
8. No active infection, including: negative HIV antibody; HBV-DNA and HCV-RNA were negative; Inactive tuberculosis There are no other active infections that require intravenous antibiotic treatment.
9. It was determined by the researchers that lymphocyte clearance therapy could be carried out.
10. If female subjects are fertile, effective contraceptive measures must be taken; Male subjects must take effective contraceptive measures during the treatment period and within 6 months after the treatment.
11. It is capable of performing normal venous blood collection and machine single blood collection, and can establish the venous access required for collection. There are no contraindications for white blood cell collection.

Exclusion Criteria:

Central nervous system (CNS) metastasis, leptomeningeal disease or metastatic central compression; 2. Have a history of bone marrow or organ transplantation; 3. There is a history of other primary malignant tumors within 5 years before the study and treatment (except for cured cervical carcinoma in situ, thyroid cancer, localized basal cell carcinoma of the skin or squamous cell carcinoma); Those with two or more malignant tumors; 4. Those who meet any of the following: A. HIV infection (positive for HIV antibody); b. Active HBV infection (HBV DNA > 500 copies /ml or 100 IU/ml); c. Active HCV infection (positive for HCV antibody, positive for HCV-RNA); d. Syphilis infected individuals (TP-Ab positive); e. Subjects with known active pulmonary tuberculosis (TB); 5. Those who are allergic to any of the drug components used in the study (including but not limited to detoxification drugs); 6. Patients who have received cell therapy previously; 7. Adverse events of previous anti-tumor treatments have not yet recovered to grade ≤1 in the CTCAE 5.0 rating before administration (except for toxicities judged by the investigator as having no safety risks, such as alopecia, pigmentation, grade 2 peripheral neurotoxicity, and stable hypothyroidism after hormone replacement therapy, etc.); 8. There was an uncontrolled active infection within 4 weeks before signing the informed consent form, and parenteral antibiotic, antiviral or antifungal treatment was required; 9. Have a history of interstitial lung disease or interstitial pneumonia, either concomitant or in the past; 10. Suffering from active or potentially recurrent autoimmune diseases; 11. Have received systemic corticosteroid (prednisone > 10mg/ day or equivalent doses of similar drugs) or other immunosuppressant therapy within 14 days prior to the first use of the study drug (except in the following circumstances: allowing local, ocular, intra-articular, intranasal and inhaled corticosteroid therapy; Short-term use of corticosteroids for preventive treatment, such as preventing contrast agent allergy; Glucocorticoid patients with physiological replacement therapy doses; 12. Abnormal laboratory tests: Absolute neutrophil count < 1.5×10^9/L; Platelet count < 75×10^9/L; Hemoglobin < 80g/ ALT or AST> 2.5×ULN; Total bilirubin > 2×ULN; Serum creatinine clearance rate < 60mL/min; 13. There was bleeding requiring medical intervention within 4 weeks before signing the informed consent form, including esophageal variceal bleeding; 14. Have received attenuated/inactivated vaccines within 4 weeks after signing the informed consent form, or plan to receive attenuated/inactivated vaccines during the screening period; Or have received attenuated/inactivated vaccines within two weeks before clearing the forest; 15. Have received anti-tumor treatments such as systemic chemotherapy, radiotherapy, targeted therapy, endocrine therapy, biological therapy and immunotherapy within 4 weeks before the first use of the study drug, except for the following: Nitrosyrea or mitomycin C within 6 weeks before the first use of the study drug; Oral fluorouracil, small molecule targeted drugs and traditional Chinese medicines with anti-tumor indications were taken within two weeks before the first use of the study drugs. Local palliative radiotherapy is within 2 weeks before the first use of the study drug; 16. Have received other unmarketed clinical research drugs or treatments within 4 weeks before the first use of the investigational drug; 17. Had undergone major organ surgery (excluding puncture biopsy diagnostic treatment) or suffered severe trauma within 4 weeks before the first use of the study drug, or required elective surgery during the trial; 18. There were severe non-healing wounds/ulcers/fractures, etc. within 4 weeks before the first use of the study drug; 19. Have a serious history of cardiovascular and cerebrovascular diseases, including but not limited to:

1. There are severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, second-to-third-degree atrioventricular block, etc.
2. Those with grade II to IV cardiac insufficiency according to the standards of the New York Heart Association (NYHA) in the United States;
3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 or above cardiovascular and cerebrovascular events occurred within 6 months before the first administration;
4. Clinically uncontrollable hypertension (blood pressure still cannot be controlled at systolic blood pressure < 140 mmHg and/or diastolic blood pressure < 90 mmHg after antihypertensive treatment);
5. Any factors that increase the risk of prolonged QTc or arrhythmia, such as heart failure, uncorrected hypokalemia, congenital long QT syndrome, or the need to use any concomitant drugs known to prolong the QT interval; 20. It is known that uveitis of grade ≥ 2 and retinopathy, etc. 21.. Known, recorded or suspected drug abuse subjects; 22. Pregnant or lactating women; 23. The researchers believe that the subjects have mental disorders, poor compliance, intolerance to apheresis, a history of other serious systemic diseases, or other reasons and are not suitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | 28 days after injection
  DLT evaluation period: The DLT evaluation period is defined as within 28 days (inclusive) after the subjects' first infusion of YC-T-001 cells during the dose escalation stage. All adverse events should be graded and evaluated in accordance with CTCAE v5.0. Among them, cytokine release syndrome (CRS) and immune effector cell-related neurotoxicity syndrome (ICANS) should be determined and graded in accordance with the standards of the American Society for Transplantation and Cell Therapy (ASTCT).
The Occurrence of Adverse Events | From the signing of the informed consent form by the subjects until within 90 days after the last injection, or when other anti-tumor treatment regimens have been initiated
  Any adverse medical event that occurs in patients or subjects of drug clinical research. It does not necessarily have a causal relationship with drug treatment or research procedures. Therefore, AE can be any adverse signs (including abnormal laboratory indicators), symptoms or diseases (new or aggravated) that are not related to the purpose of medication and have a temporal correlation with the investigational drug, regardless of whether these situations have a causal relationship with the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, The First Affiliated Hospital of Jilin University, Changchun, Jilin, China